CLINICAL TRIAL: NCT00287950
Title: Protocol for Infants With Neuroblastoma Diagnosed Under the Age of One Year
Brief Title: Combination Chemotherapy, Surgery, and Radiation Therapy in Treating Infants With Neuroblastoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454726; CCLG-1992-05; EU-20593; CCLG-9205
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2006-12

CONDITIONS: Neuroblastoma
Keywords: disseminated neuroblastoma; localized resectable neuroblastoma; localized unresectable neuroblastoma; regional neuroblastoma; stage 4S neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Carboplatin; Cisplatin; Cyclophosphamide; Etoposide; Vincristine; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: etoposide
Drug: vincristine sulfate
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving chemotherapy and radiation therapy after surgery may kill any tumor cells that remain after surgery. Sometimes, the tumor may not need any treatment until it progresses. In this case, observation may be sufficient.

PURPOSE: This clinical trial is studying how well giving combination chemotherapy together with surgery and radiation therapy works in treating infants with neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Register all children < 12 months of age diagnosed with neuroblastoma.
* Evaluate possible prognostic factors in these patients with particular reference to the collection of biological material.
* Correlate outcome with factors other than stage in these patients.
* Determine criteria to modify treatment for some children with advanced disease without impairing survival.

OUTLINE: This is a nonrandomized, multicenter study. Patients are assigned to 1 of 4 treatment groups according to disease stage.

* Group 1 (stage 1, 2A, or 2B disease): Patients undergo surgical resection of the tumor. Patients with paraspinal tumors may receive chemotherapy* to shrink the tumor before undergoing surgery. Patients with local recurrence after surgery proceed to treatment as in group 3. Patients with metastatic recurrence after surgery proceed to treatment as in group 4.
* Group 2 (stage 4S disease): Patients undergo observation only. Patients with hepatomegaly or progressive disease may receive chemotherapy*. Patients who do not respond to chemotherapy may undergo up to 4 courses of radiotherapy.
* Group 3 (stage 3 disease): Patients receive OPEC chemotherapy comprising vincristine IV and cyclophosphamide IV on day 1, cisplatin IV continuously over 24 hours on day 1, and etoposide IV over 4 hours on day 3 during courses 1, 3, and 5. Patients receive OJEC chemotherapy comprising vincristine IV, cyclophosphamide IV, etoposide IV over 4 hours, and carboplatin IV over 1 hour on day 1 during courses 2, 4, and 6. Courses repeat every 3 weeks with alternating OPEC and OJEC chemotherapy for 6 courses. Patients with residual disease then receive 4 additional courses of alternating OPEC and OJEC chemotherapy. Patients whose tumor becomes resectable after either 6 or 10 courses of chemotherapy undergo surgery. Patients with residual disease after 10 courses of chemotherapy are assessed by regular scans. Patients with disease progression on scans undergo radiotherapy. Patients with ganglioneuroma or total necrosis only with no evidence of neuroblastoma after either 6 or 10 courses of chemotherapy receive no further treatment.
* Group 4 (stage 4 disease): Patients receive alternating courses of OPEC and OJEC for 6 courses as in group 3. Patients who do not achieve metastatic complete response (CR) receive 4 additional courses of alternating OPEC and OJEC chemotherapy. Patients achieving metastatic CR after either 6 or 10 courses of chemotherapy undergo surgery to remove the tumor. Patients with macroscopic residual disease on resected specimen receive 4 additional courses of alternating OPEC and OJEC chemotherapy and then undergo biopsy. Patients with residual disease on biopsy are assessed by regular scans. Patients with disease progression on scans undergo radiotherapy. Patients with ganglioneuroma or total necrosis only after surgery with or without the 4 additional courses of chemotherapy receive no further treatment.

NOTE: * OJEC chemotherapy with a lower dose of carboplatin

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 120 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed newly diagnosed neuroblastoma

  * Any stage disease
  * No previously treated disease
  * Must be diagnosed before the first birthday
* Must be able to start treatment before reaching 13 months of age

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 1992-09

CONTACTS AND LOCATIONS:
Overall Officials: Penelope Brock, MD, PhD, Study Chair — University College London Hospitals; Mary P. Gerrard, MBChB, FRCP, FRCPCH — Children's Hospital - Sheffield; Andrew David J. Pearson, MD, FRCP, DCh — University of Newcastle Upon-Tyne; S. J. Keith Holmes, DO — St. George's Hospital; Ann Barrett — University of Glasgow
Locations (22):
- Our Lady's Hospital for Sick Children, Dublin, Ireland
- United Kingdom (21):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Royal London Hospital, London, England
  - Great Ormond Street Hospital for Children NHS Trust, London, England
  - Meyerstein Institute of Oncology at University College of London Hospitals, London, England
  - Central Manchester and Manchester Children's University Hospitals NHS Trust, Manchester, England
  - Sir James Spence Institute of Child Health, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales